CLINICAL TRIAL: NCT04861584
Title: Phase II Study of Neoadjuvant Toripalimab with Gemcitabine-Cisplatin in Subjects with T2-4aN0M0 Bladder Cancer: GZZJU-2021NB
Brief Title: Neoadjuvant Toripalimab in Combination with Gemcitabine and Cisplatin Therapy in Local Advanced Bladder Cancer Subjects
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Abai Xu, Vice Director, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZZJU-2021NB
Record Dates: First submitted 2021-04-09; First posted 2021-04-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-03

CONDITIONS: Urinary Bladder Cancer
Keywords: bladder cancer; checkpoint inhibitor; neoadjuvant therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab+Gemcitabine/Cisplantin（GC） (Experimental): Subjects receive gemcitabine/cisplatin every 21 days, repeated for 4 cycles. . Toripalimab is given every 21 days for 4 doses starting C1D1. Subjects will then have consolidative surgery to remove their primary tumor within 6 weeks after their last dose of neoadjuvant therapy.
  Interventions: Drug: Neoadjuvant Toripalimab in Combination With Gemcitabine and Cisplatin

INTERVENTIONS:
Drug: Neoadjuvant Toripalimab in Combination With Gemcitabine and Cisplatin — 4 cycle neoadjuvant therapy and radical cystectomy
  Other Names: Toripalimab

SUMMARY:
This is a pre-surgical study involving subjects with local advanced bladder cancer, who are candidates for neoadjuvant therapy. It is a single-arm phase II portion.

DETAILED DESCRIPTION:
Outline: This study is a single-arm, open, exploratory clinical trial;

Subjects receive: gemcitabine 1000mg/m2 IV Day1 and Day8 every 21 days repeated for 4 cycles; cisplatin 35mg/m2 IV Day1 and Day2 every 21 days, repeated for 4 cycles.

Toripalimab at recommended phase II dose is given every 3 weeks for 4 doses starting with Cycle1 Day1(C1D1).

Subjects will then have surgery to remove their primary tumor within 6 weeks after their last dose of neoadjuvant therapy.

Eastern Cooperative Oncology Group (ECOG) performance status: 0-1

Demonstrate adequate organ function as defined by the following laboratory values at study entry. All screening labs should be performed within 28 days of C1D1.

Hematopoetic:

Absolute neutrophil count (ANC) ≥1,500 /mcL Absolute lymphocyte count ≥350 mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L

Renal: Measured or calculated creatinine clearance ≥30 mL/min

Hepatic:

Serum total bilirubin ≤ 1.25 X ULN OR ≤ 2.5 x ULN for subjects with Gilbert's disease Aspartate aminotransferase (AST, SGOT) and alanine aminotransferase (ALT, SGPT) ≤ 2 X ULN

Coagulation:

International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy and as long as PT or PTT is within therapeutic range of intended use of anticoagulants

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years old on day of signing informed consent, regardless of gender;
* ECOG score 0-1 points, expected survival time> 6 months;
* Pathologically confirmed locally advanced bladder urothelial carcinoma (cT2-T4a, N≤1, M0, tumor staging according to American Joint Committee on Cancer (AJCC), 2017, eighth edition);
* Appropriate and plan for radical cystectomy;
* According to the RECIST1.1 standard, there is at least one measurable lesion (spiral CT scan ≥10mm);
* Since the diagnosis of locally advanced bladder urothelial carcinoma, patient has not received anti-tumor system treatment;
* The main organ functions are normal, and the following requirements must be met within 2 weeks before the first study treatment:
* Routine blood examination must meet: WBC≥4.0×109/L; PLT≥90×109/L; Hb≥90g/L (patients can be infused with red blood cells to meet this standard);
* Blood biochemical examination must meet: serum creatinine (Cr) ≤1.5 times the upper limit of normal (ULN) or endogenous creatinine clearance ≥60mL/min; TBIL≤1.5×ULN; ALB≥30g/L; ALT and AST≤ 3.0×ULN; TSH≤1.5×ULN.
* Female patients with fertility must undergo a pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and they voluntarily adopt appropriate methods of contraception during the observation period and within 8 weeks after the last administration;
* Agree to provide diagnosis and treatment-related tumor tissue specimens for clinical research, and have the ability to follow the planned research visit until the clinical recurrence/progress is clear.
* Sign informed consent voluntarily.

Exclusion Criteria:

* Have previously received anti-PD1/PDL1/CTLA-4 antibody treatment or systemic chemotherapy, bladder infusion chemotherapy is excluded;
* Have received bladder bacille Calmette Guerin (BCG) infusion therapy within 4 weeks;
* Have received radiotherapy of the bladder in the past;
* Patients with any history of active autoimmune disease or autoimmune disease;
* Complicated diseases that require the use of immunosuppressive drugs; concurrent diseases that require the use of immunosuppressive agents for systemic or locally absorbable corticosteroids. It is forbidden to use prednisone greater than 10 mg/day or the same dose in the 2 weeks before the use of the study drug;
* Combined with other malignant tumors;
* Have a history of allergy to other antibody drugs;
* The history of human immunodeficiency virus (HIV) infection;
* The subject has active infection, including active tuberculosis;
* Combined with severe heart disease, or combined with New York Heart Association (NYHA) grade 3 or 4 cardiac insufficiency;
* Kidney transplant patients;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2026-10-03 (Estimated); Study Completion 2027-04-03 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate evaluated after 4 cycles of neoadjuvant Toripalimab in combination with gemcitabine and cisplatin at time of radical cystectomy, each cycle is 21 days | Up to 90 days after last dose of investigation product
  the absence of residual muscle invasive bladder cancer in surgical specimens of cystectomy (pathologically decreased to ≤pT1N0, including pT0, pT1, pTa and pTis

SECONDARY OUTCOMES:
Safety assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4 criteria | From the first day of the treatment to the end of neoadjuvant treatment, assessed up to 6 month
  To assess safety of Toripalimab in combination with gemcitabine and cisplatin in patients with bladder cancer according to CTCAE v4 criteria
Progression-free survival assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 | From the start of neoadjuvant therapy to the time when any disease progression is first recorded. Assessed lasted for 24 months, calculated from the date of enrolled
  From the start of neoadjuvant therapy to the time when any disease progression is first recorded, disease progression includes the progression detected by clinical or imaging before cystectomy, as well as the distant metastasis or pelvic recurrence after cystectomy. Newly discovered primary tumors in other parts of the urinary tract such as renal pelvis, ureter and urethra are not considered as disease progression.
Tumor immune microenvironment indicators assessed by Microenvironment Analysis Panel | Assessed lasted for 24 months, calculated from the date of enrolled
  The expression rate of PDL1 in pathological specimens assessed by Burning Rock's product OncoScreen plus+Microenvironment Analysis Panel at the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Abai Xu, doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China